CLINICAL TRIAL: NCT02167139
Title: A Randomised, Double-blind, Parallel Group, Multicentre Clinical Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Immunogenicity of SB5 Compared to Humira® in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study Comparing SB5 to Humira® in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB5-G31-RA
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB5 (proposed biosimilar to adalimumab) (Experimental): SB5 40 mg every other week via subcutaneous injection
  Interventions: Drug: SB5 (proposed biosimilar to adalimumab)
- Humira (adalimumab) (Active Comparator): Humira 40 mg every other week via subcutaneous injection
  Interventions: Drug: Humira (adalimumab); Drug: SB5 (proposed biosimilar to adalimumab)

INTERVENTIONS:
Drug: Humira (adalimumab)
  Arms: Humira (adalimumab)
Drug: SB5 (proposed biosimilar to adalimumab)

SUMMARY:
This is a randomised, double-blind, parallel group, multicentre clinical study to evaluate the efficacy, safety, tolerability, pharmacokinetics and immunogenicity of SB5 compared to Humira® in subjects with moderate to severe RA despite MTX therapy.

DETAILED DESCRIPTION:
Investigational product: SB5 40 mg (0.8 mL of 50 mg/mL) Indication studied: Rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Are male or female aged 18-75 years at the time of signing the informed consent form.
* Have been diagnosed as having RA according to the revised 1987 American College of Rheumatology (ACR) criteria for at least 6 months but not exceeding 15 years prior to Screening.
* Have moderate to severe active disease despite MTX therapy defined as:

  1. More than or equal to six swollen joints and more than or equal to six tender joints (from the 66/68 joint count system) at Screening and Randomisation.
  2. Either erythrocyte sedimentation rate (Westergren) ≥ 28 mm/h or serum C-reactive protein ≥ 10 mg/dL at Screening.
* Must have been treated with MTX for a total of at least 6 months prior to Randomisation and must have been on both: a stable route of administration (oral or parenteral) and stable dose of MTX (10-25 mg/week) for at least 4 weeks prior to Screening.
* Female subjects who are not pregnant or nursing at Screening and Randomisation and who are not planning to become pregnant from Screening until 5 months after the last dose of IP.

Exclusion Criteria:

* Have been treated previously with any biological agents including any tumour necrosis factor inhibitor.
* Have a known hypersensitivity to human immunoglobulin proteins or other components of Humira or SB5.
* Have a positive serological test for hepatitis B or hepatitis C or have a known history of infection with human immunodeficiency virus.
* Have a current diagnosis of active tuberculosis (TB), have been recently exposed to a person with active TB, or are considered to have latent TB.
* Have had a serious infection or have been treated with intravenous antibiotics for an infection within 8 weeks or oral antibiotics within 2 weeks prior to Randomisation.
* Have a history of chronic or recurrent infection.
* Have any of the following conditions:

  1. History of congestive heart failure (New York Heart Association Class III/IV).
  2. History of acute myocardial infarction or unstable angina within the previous 12 months prior to Screening.
  3. History of demyelinating disorders.
  4. History of any malignancy within the previous 5 years prior to Screening.
  5. History of lymphoproliferative disease including lymphoma.
  6. Any other disease or disorder which, in the opinion of the Investigator, will put the subject at risk if they are enrolled.
* Have physical incapacitation (ACR functional Class IV or wheelchair-/bed-bound).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asta Baranauskaite, M.D., Ph.D., Principal Investigator — Hospital of Lithuanian University of Health Sciences
Locations (2):
- Investigational Site, Kaunas, Lithuania
- Investigational site, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Emery P, Suh CH, Weinblatt ME, Smolen JS, Keystone EC, Genovese M, Vencovsky J, Kay J, Hong E, Baek Y, Ghil J. Impact of immunogenicity on efficacy and tolerability of tumour necrosis factor inhibitors: pooled analysis of biosimilar studies in rheumatoid arthritis. Scand J Rheumatol. 2020 Sep;49(5):361-370. doi: 10.1080/03009742.2020.1732458. Epub 2020 May 29. PMID 32468892
- [Derived] Smolen JS, Choe JY, Weinblatt ME, Emery P, Keystone E, Genovese MC, Myung G, Hong E, Baek I, Ghil J. Pooled analysis of TNF inhibitor biosimilar studies comparing radiographic progression by disease activity states in rheumatoid arthritis. RMD Open. 2020 Jan;6(1):e001096. doi: 10.1136/rmdopen-2019-001096. PMID 31958281
- [Derived] Weinblatt ME, Baranauskaite A, Dokoupilova E, Zielinska A, Jaworski J, Racewicz A, Pileckyte M, Jedrychowicz-Rosiak K, Baek I, Ghil J. Switching From Reference Adalimumab to SB5 (Adalimumab Biosimilar) in Patients With Rheumatoid Arthritis: Fifty-Two-Week Phase III Randomized Study Results. Arthritis Rheumatol. 2018 Jun;70(6):832-840. doi: 10.1002/art.40444. Epub 2018 Apr 24. PMID 29439289
- [Derived] Weinblatt ME, Baranauskaite A, Niebrzydowski J, Dokoupilova E, Zielinska A, Jaworski J, Racewicz A, Pileckyte M, Jedrychowicz-Rosiak K, Cheong SY, Ghil J. Phase III Randomized Study of SB5, an Adalimumab Biosimilar, Versus Reference Adalimumab in Patients With Moderate-to-Severe Rheumatoid Arthritis. Arthritis Rheumatol. 2018 Jan;70(1):40-48. doi: 10.1002/art.40336. Epub 2017 Nov 21. PMID 28950421

RESULTS

PARTICIPANT FLOW:
Groups:
- SB5 (Proposed Biosimilar to Adalimumab): SB5 40 mg every other week via subcutaneous injection SB5 (proposed biosimilar to adalimumab)
- Humira (Adalimumab): Humira 40 mg every other week via subcutaneous injection to Week 24, then randomised again in a 1:1 ratio to either continue on Humira® 40 mg (Humira®/Humira®) or be transitioned to SB5 40 mg (Humira®/SB5) every other week up to Week 50.
- Humira (Adalimumab), Switch to SB5: From Week 24, SB5 40 mg (Humira®/SB5) every other week up to Week 50.
- Humira (Adalimumab), Continue as Humira: From Week 24, Humira® 40 mg (Humira®/Humira®) every other week up to Week 50.
Period: Randomised, Double-blind
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab) | Humira (Adalimumab), Switch to SB5 | Humira (Adalimumab), Continue as Humira
Started | 271 | 273 | 0 | 0
Completed | 254 | 254 | 0 | 0
Not Completed | 17 | 19 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 8 | 0 | 0
Not completed — Adverse Event | 2 | 9 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0
Period: Transition-extension
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab) | Humira (Adalimumab), Switch to SB5 | Humira (Adalimumab), Continue as Humira
Started | 254 | 0 | 125 | 129
Completed | 248 | 0 | 117 | 124
Not Completed | 6 | 0 | 8 | 5
Not completed — Adverse Event | 2 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 4 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Humira (Adalimumab): Humira 40 mg every other week via subcutaneous injection
  Humira (adalimumab)
  SB5 (proposed biosimilar to adalimumab)
- Total: Total of all reporting groups
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab) | Total
Number analyzed (Participants) | 271 | 273 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.67) | 52.5 (11.91) | 51.2 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 224 | 441
  Male | 54 | 49 | 103

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% Response Criteria (ACR20)
Time Frame: Week 24
Measure: Number; unit: percentage of participants
Groups:
- SB5 (Proposed Biosimilar to Adalimumab): SB5 40 mg every other week via subcutaneous injection up to Week 24
- Humira (Adalimumab): Humira 40 mg every other week via subcutaneous injection up to Week 24
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab)
Number analyzed (Participants) | 239 | 237
percentage of participants | 72.4 | 72.2

2. Secondary Outcome: ACR20
Time Frame: Week 52
Measure: Number; unit: percentage of participants
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab), Switch to SB5 | Humira (Adalimumab), Continue as Humira
Number analyzed (Participants) | 212 | 106 | 111
percentage of participants | 76.9 | 81.1 | 71.2

3. Secondary Outcome: American College of Rheumatology 50% Response Criteria (ACR50)
Time Frame: Week 24, Week 52
Measure: Number; unit: percentage of participants
Groups:
- SB5 (Proposed Biosimilar to Adalimumab) at Week 24; SB5 (Proposed Biosimilar to Adalimumab) at Week 52: SB5 40 mg every other week via subcutaneous injection SB5 (proposed biosimilar to adalimumab)
- Humira (Adalimumab) at Week 24: Humira 40 mg every other week via subcutaneous injection to Week 24, then randomised again in a 1:1 ratio to either continue on Humira® 40 mg (Humira®/Humira®) or be transitioned to SB5 40 mg (Humira®/SB5) every other week up to Week 50.
- Humira (Adalimumab), Switch to SB5 at Week 52: From Week 24, SB5 40 mg (Humira®/SB5) every other week up to Week 50.
- Humira (Adalimumab), Continue as Humira at Week 52: From Week 24, Humira® 40 mg (Humira®/Humira®) every other week up to Week 50.
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) at Week 24 | Humira (Adalimumab) at Week 24 | SB5 (Proposed Biosimilar to Adalimumab) at Week 52 | Humira (Adalimumab), Switch to SB5 at Week 52 | Humira (Adalimumab), Continue as Humira at Week 52
Number analyzed (Participants) | 239 | 237 | 212 | 106 | 111
percentage of participants | 38.1 | 39.7 | 49.1 | 53.8 | 51.4

4. Secondary Outcome: Disease Activity Score Based on a 28 Joint Count (DAS28)
Time Frame: Week 24, Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SB5 (Proposed Biosimilar to Adalimumab) | Humira (Adalimumab)
All-Cause Mortality (participants affected / at risk) | 0/268 | 0/273
Serious Adverse Events (participants affected / at risk) | 9/268 | 16/273
Other Adverse Events (participants affected / at risk) | 35/268 | 44/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB5 (Proposed Biosimilar to Adalimumab) (N=268) | Humira (Adalimumab) (N=273)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lumber radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB5 (Proposed Biosimilar to Adalimumab) (N=268) | Humira (Adalimumab) (N=273)
Nasopharyngitis (Infections and infestations) | 24 (27) | 30 (34)
Headache (Nervous system disorders) | 11 (13) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow Sponsor sixty (60) days to review and comment on them.